CLINICAL TRIAL: NCT00004390
Title: Phase III Randomized Controlled Study of Morphine and Nortriptyline in the Management of Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Johns Hopkins University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 199/12133; JHUSM-93010802
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-02

CONDITIONS: Pain; Herpes Zoster
Keywords: disease-related problem/condition; herpes zoster infection; herpesvirus infection; immunologic disorders and infectious disorders; pain; rare disease; viral infection
MeSH Terms: conditions — Pain; Herpes Zoster; Chickenpox; Herpesviridae Infections; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Desipramine; Methadone; Morphine; Nortriptyline

INTERVENTIONS:
Drug: desipramine
Drug: methadone
Drug: morphine
Drug: nortriptyline

SUMMARY:
OBJECTIVES: I. Determine whether opioid (morphine) treatment results in better management of pain than treatment with tricyclic antidepressant (nortriptyline).

II. Assess the effects the two treatments have on affective and cognitive functions.

III. Determine whether the presence of psychiatric comorbidity, particularly depression, can predict the outcome of the two treatments.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, crossover study. Patients are stratified by the duration of pain (greater than 1 year or no greater than 1 year) and the presence or absence of major depression.

Patients are randomized into 6 treatment order groups. Patients start with nortriptyline, morphine, or placebo, taken orally every day. If patients are unable to tolerate nortriptyline or morphine, they will receive desipramine or methadone instead.

A drug titration period lasting 3 weeks is ensued for administration of the first drug treatment. The goal of this titration period is to gradually increase the dose of the drug to obtain maximal analgesic efficacy. Drug dosage is maintained for a period of 3 weeks. The drug dosage is tapered off and followed by a drug free period of 1 week.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnostically confirmed postherpetic neuralgia for at least 3 months following a segmental herpes zoster eruption

--Prior/Concurrent Therapy--

* Other: No concurrent monoamine oxidase inhibitors

--Patient Characteristics--

* Life expectancy: At least 6 months
* Cardiovascular: No second degree or complete heart blockage No myocardial infarction in the last 3 months
* Pulmonary: No severe pulmonary disease
* Other: No history of substance abuse No history of dementia No history of encephalopathy No severe depression that precludes withdrawal from antidepressants Not pregnant No angle-closure glaucoma No AIDS related disease complex No terminal disease with life expectancy of less that 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1995-02

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasa N. Raja, Study Chair — Johns Hopkins University